CLINICAL TRIAL: NCT02743702
Title: Effectiveness of a Protocol of Respiratory Physiotherapy for Improvement or Maintenance of Respiratory Function, and Incidence of Respiratory Infections in Children With Neuromuscular Diseases, Compared With no Approach by Respiratory Physiotherapy of Respiratory Difficulties: A Randomized Clinical Trial With Two Groups in Parallel With Blinded Evaluator.
Brief Title: Effectiveness of Respiratory Physiotherapy in Children With Neuromuscular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, JJ JIMENEZ-REJANO, PhD, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USeville-JJIMENEZ-REJANO
Record Dates: First submitted 2016-04-05; First posted 2016-04-19 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Neuromuscular Diseases
Keywords: Effectiveness; Physical therapy modalities; neuromuscular diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- GROUP RECEIVING RESPIRATORY PHYSIOTHERAPY (Experimental): Respiratory Physiotherapy sessions were held once a week by the physiotherapist, and four times more for the family at home, for one year. The sessions have a duration between 30 and 45 minutes, varying according to the level of patient cooperation. The exercise program should be repeated in three cycles, although younger children took longer than older in performing them.
  Interventions: Other: RESPIRATORY PHYSIOTHERAPY; Other: USUAL THERAPIES
- GROUP RECEIVING THEIR USUAL THERAPIES (Experimental): This group received no approach of their respiratory difficulties by Physiotherapy. Only continued their usual therapies.
  Interventions: Other: USUAL THERAPIES

INTERVENTIONS:
Other: RESPIRATORY PHYSIOTHERAPY — The protocol designed was composed of the following exercises:
  * supine position: inhalation and exhalation with abdominal and thoracic pressures. 5 times
  * lateral decubitus, with incentive spirometer lung inflation are made on right/left sides. 3 sets on each side
  * sitting position, with the body leaning slightly forward, head and shoulders bent inwardly directed. It inspire called for 3 times, sent off in air through the mouth, after that the child was coughing
  * diaphragmatic breathing in a sitting position: after a slow exhalation requested, child should steam a mirror with his mouth slightly open. 3 replications
  * in a sitting position, with help of an ambu bag, we made inflations. Repeated 3 times
  * exercises of upper member coupled to respiratory rhythm: shoulder flexion and extension was carried out during the inspiratory phase and the extension and adduction of them during expiration. 3 times
  Arms: GROUP RECEIVING RESPIRATORY PHYSIOTHERAPY
Other: USUAL THERAPIES

SUMMARY:
The main objective of this study is to determine whether the Respiratory Physiotherapy allows improvement or maintenance of respiratory function in children with Neuromuscular Diseases, against respiratory deterioration that occurs in the group of subjects who did not receive this treatment. And to determine whether decreasing the number of respiratory infections and secondly the need for antibiotics and the number of emergency room visits and hospital admissions related to these.

DETAILED DESCRIPTION:
Background:

Many authors have demonstrated the efficacy of Physiotherapy in Respiratory attending respiratory difficulties associated with different types of pathologies (Chronic Obstructive Pulmonary Disease, cystic fibrosis, tumors), however the investigators did not find studies with scientific evidence demonstrating the effectiveness of these programs in children with Neuromuscular Diseases (NMD), whose quality and life expectancy depends largely on the proper handling of Bronchial secretions and delay the deterioration of respiratory function.

The main objective of this study focuses on determining the effectiveness of physiotherapy for the treatment of respiratory breathing difficulties in children with NMD. Deducing other aspects such as the impact of this program on the number of visits to hospital emergencies department each year, hospital admissions and respiratory infections suffered by these children, and the need or not of antibiotics.

Material and method:

This research is an analytical, longitudinal, prospective, experimental, evaluator blinded study. It is controlled with two parallel groups, randomized clinical trial.

The sample consisted of children diagnosed with NMD. For the evolution of different variables spirometric test was used for variables related to the function respiratory, and a tracking sheet designed by the researchers to collect the number hospital emergency visits each year, as well as hospital admissions, respiratory infections and need of antibiotics. These assessments were made before and after the start of program and during every four months.

Patients were randomized to control or experimental group, no apply any Respiratory Physical Therapy treatment in subjects in the first group and performing a Respiratory Physical Therapy program in the second. This program was carried out once in week by the physiotherapist, and four times weekly at home, by family, during one year.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with a Disease of the Neuromuscular junction, according to International Classification of Diseases 10.
* Be aged between 3 and 18 years.

Exclusion Criteria:

* Being unable to perform spirometry, for physical or psychological difficulties.
* Be involved in another program Respiratory Physiotherapy.
* Present some kind of associated pathology (such as broken ribs, state epilepticus ...) in which it is contraindicated any maneuvers of the respiratory therapy protocol designed.
* If researchers are informed of the existence of a serious illness of the father / mother / tutor that preclude to carrying out the program of respiratory Physiotherapy at home.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo de Investigación Área de Fisioterapia CTS 305 - Universidad de Sevilla, Seville, Sevilla, Spain

REFERENCES:
- [Background] Ambrosino N, Vitacca M, Rampulla C. Standards for rehabilitative strategies in respiratory diseases. Monaldi Arch Chest Dis. 1995 Aug;50(4):293-318. No abstract available. PMID 7550210
- [Background] Danov Z, Schroth MK. Respiratory management of pediatric patients with neuromuscular disease. Pediatr Ann. 2010 Dec;39(12):769-76. doi: 10.3928/00904481-20101116-07. No abstract available. PMID 21162485
- [Background] Bach JR, Ishikawa Y, Kim H. Prevention of pulmonary morbidity for patients with Duchenne muscular dystrophy. Chest. 1997 Oct;112(4):1024-8. doi: 10.1378/chest.112.4.1024. PMID 9377912
- [Background] Chatwin M, Ross E, Hart N, Nickol AH, Polkey MI, Simonds AK. Cough augmentation with mechanical insufflation/exsufflation in patients with neuromuscular weakness. Eur Respir J. 2003 Mar;21(3):502-8. doi: 10.1183/09031936.03.00048102. PMID 12662009
- [Background] Vianello A, Corrado A, Arcaro G, Gallan F, Ori C, Minuzzo M, Bevilacqua M. Mechanical insufflation-exsufflation improves outcomes for neuromuscular disease patients with respiratory tract infections. Am J Phys Med Rehabil. 2005 Feb;84(2):83-8; discussion 89-91. doi: 10.1097/01.phm.0000151941.97266.96. PMID 15668554
- [Background] Watzek I, Winterholler M. [Basic principles of non-respiratory physiotherapy for neuromuscular diseases]. Pneumologie. 2008 Mar;62 Suppl 1:S28-30. doi: 10.1055/s-2007-1016426. German. PMID 18317980

RESULTS

PARTICIPANT FLOW:
Groups:
- GROUP RECEIVING RESPIRATORY PHYSIOTHERAPY: Respiratory Physiotherapy sessions were held once a week by the physiotherapist, and four times more for the family at home, for one year. The sessions have a duration between 30-45 minutes, varying according to the level of patient cooperation. The exercise program should be repeated in three cycles, although younger children took longer than older in performing them.
  RESPIRATORY PHYSIOTHERAPY: The protocol designed was composed of the following exercises:
  * supine position: inhalation and exhalation with abdominal and thoracic pressures. 5 times
  * lateral decubitus, with incentive spirometer lung inflation are made on right/left sides. 3 sets on each side
  * sitting position, with the body leaning slightly forward, head and shoulders bent inwardly directed. It inspire called for 3 times, sent off in air through the mouth, after that the child was coughing
  * diaphragmatic breathing in a sitting position: after a slow exhalation requested, child should steam a mirror with his
- GROUP RECEIVING THEIR USUAL THERAPIES: This group received no approach of their respiratory difficulties by Physiotherapy. Only continued their usual therapies.
  USUAL THERAPIES
Period: Overall Study
Arm/Group | GROUP RECEIVING RESPIRATORY PHYSIOTHERAPY | GROUP RECEIVING THEIR USUAL THERAPIES
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GROUP RECEIVING RESPIRATORY PHYSIOTHERAPY | GROUP RECEIVING THEIR USUAL THERAPIES | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6 [4 to 9] | 7.5 [3.75 to 9.25] | 7 [4 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Vital Capacity at One Year.
Description: Change from Baseline vital capacity at one year evaluated by spirometer.
Time Frame: At baseline and at 1 year
Measure: Median (Inter-Quartile Range); unit: percentage of Change of vital capacity
Groups:
- GROUP RECEIVING RESPIRATORY PHYSIOTHERAPY: Respiratory Physiotherapy sessions were held once a week by the physiotherapist, and four times more for the family at home, for one year. Sessions have a duration between 30-45 minutes, varying according to the level of patient cooperation. The exercise program should be repeated in three cycles, although younger children took longer than older in performing them.
  RESPIRATORY PHYSIOTHERAPY: The protocol designed was composed of the following exercises:
  * supine position: inhalation and exhalation with abdominal and thoracic pressures. 5 times
  * lateral decubitus, with incentive spirometer lung inflation are made on right/left sides. 3 sets on each side
  * sitting position, with the body leaning slightly forward, head and shoulders bent inwardly directed. It inspire called for 3 times, sent off in air through the mouth, after that the child was coughing
  * diaphragmatic breathing in a sitting position: after a slow exhalation requested, child should steam a mirror with his mou
Arm/Group | GROUP RECEIVING RESPIRATORY PHYSIOTHERAPY | GROUP RECEIVING THEIR USUAL THERAPIES
Number analyzed (Participants) | 11 | 10
percentage of Change of vital capacity | 33.33 [11.11 to 89.74] | -7.41 [-15.60 to -3.82]
Statistical Analysis 1: Comparison: GROUP RECEIVING RESPIRATORY PHYSIOTHERAPY vs GROUP RECEIVING THEIR USUAL THERAPIES; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- GROUP RECEIVING RESPIRATORY PHYSIOTHERAPY: Respiratory Physiotherapy sessions were held once a week by the physiotherapist, and four times more for the family at home, for 1 year. The sessions have a duration between 30-45 minutes, varying according to the level of patient cooperation. The exercise program should be repeated in three cycles, although younger children took longer than older in performing them.
  RESPIRATORY PHYSIOTHERAPY: The protocol designed was composed of the following exercises:
  * supine position: inhalation and exhalation with abdominal and thoracic pressures. 5 times
  * lateral decubitus, with incentive spirometer lung inflation are made on right/left sides. 3 sets on each side
  * sitting position, with the body leaning slightly forward, head and shoulders bent inwardly directed. It inspire called for 3 times, sent off in air through the mouth, after that the child was coughing
  * diaphragmatic breathing in a sitting position: after a slow exhalation requested, child should steam a mirror with his mou
Arm/Group | GROUP RECEIVING RESPIRATORY PHYSIOTHERAPY | GROUP RECEIVING THEIR USUAL THERAPIES
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes